CLINICAL TRIAL: NCT06203392
Title: Effects of a Very Low Carbohydrate Ketogenic Diet Versus Mediterranean Diet on Markers of Bone Health and Muscle Function in Older Adults: A Pilot Study
Brief Title: Effects of a Very Low Carbohydrate Ketogenic Diet or Mediterranean Diet on Markers of Musculoskeletal Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202301329; 2P30AG028740-16 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2024-01-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Aging; Musculoskeletal Diseases
Keywords: diet, aging, ketogenic, ketosis, Mediterranean
MeSH Terms: conditions — Musculoskeletal Diseases; Ketosis | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment of some but not all outcomes will be masked. More specifically, assessment of all outcomes determined by laboratory assay will be masked (e.g., bone turnover markers and 24-hour urine analytes).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low carbohydrate ketogenic diet for six weeks (Experimental)
  Interventions: Other: Very low carbohydrate ketogenic diet
- Mediterranean diet for six weeks (Active Comparator)
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Very low carbohydrate ketogenic diet — Very low carbohydrate ketogenic diet provided for six weeks
  Arms: Very low carbohydrate ketogenic diet for six weeks
Other: Mediterranean diet — Mediterranean diet provided for six weeks
  Arms: Mediterranean diet for six weeks

SUMMARY:
Preclinical data indicate that very low carbohydrate ketogenic diets (KD) may prevent progression of age-related sarcopenia (skeletal muscle decline) but also may disturb bone metabolism. The investigators will pilot test a randomized trial comparing the effects of short-term adaptation to a well-formulated ketogenic diet and Mediterranean diet on markers of bone metabolism and muscle function in older adults. The expected results will help inform the benefit-risk assessment for older patients considering longer term use of KD therapy.

DETAILED DESCRIPTION:
Eucaloric very low carbohydrate ketogenic diets (KD) are therapeutic diets that mimic fasting by generating ketones for metabolic fuel while meeting nutritional requirements (nutritional ketosis). Nutritional ketosis may broadly benefit healthspan through mechanisms such as suppression of inflammation or induction of autophagy, and preclinical and emerging clinical data indicate that KD therapy may help slow progression of age-related conditions including sarcopenia. However, questions remain about the benefits and risks of KD, especially relative to recommended therapeutic diets such as the Mediterranean Diet (MD) for which there is evidence of benefit for age-related conditions. For example, KD has shown efficacy for weight loss, which could reduce ectopic lipid accumulation that weakens muscle and bone. KD has been shown to increase skeletal muscle mitochondrial mass, mitochondrial activity, and strength in aged mice, possibly by increasing peroxisome proliferator-activated receptor activity and preserving fast-oxidative fibers that typically decline with age. However, long term use of KD may adversely impact bone. KD can cause deterioration of bone in juvenile mice without evidence of undernutrition and is associated with skeletal demineralization in children being treated for drug-resistant epilepsy.

Given the burden of musculoskeletal disease in older Americans, it is vital to understand the effects of KD on the musculoskeletal system of older adults to inform the benefit-risk assessment for an older patient and to optimize the effectiveness of KD for age-related conditions. The investigators are conducting a pilot test of a randomized clinical trial comparing the effects of short-term adaptation to a well-formulated KD and MD on markers of bone health and muscle function in older adults. The investigators will supply fresh prepared meals to achieve high adherence to the dietary interventions and adequate contrast in metabolic state between treatment groups.

Potential participants will complete a screening process so the investigators can determine whether potential participants are eligible to enroll in the study. At the first screening visit, the study team will measure blood pressure, height, and weight. Individuals will complete questionnaires that collect information about their health history, dietary intake, and physical activity habits. No more than 50 mL of blood will be collected from potential participants to run routine clinical lab tests to evaluate health status.

If an individual remains eligible after the first screening visit, they will be invited to complete a 24-hour urine collection (at home) and to schedule a second screening visit. At the second screening visit, a physician will conduct a physical exam and assess their body composition with an x-ray technology called dual-energy x-ray absorptiometry (DEXA or DXA).

If an individual remains eligible after the second screening visit, they will be invited to enroll in the dietary intervention study. Once enrolled, the participant will be assigned to either a very low carbohydrate ketogenic dietary pattern or a Mediterranean dietary pattern. The investigators will provide most of the food the participant will need each day in the form of a nutrition shake (breakfast) and two prepared meals (lunch and dinner). A study dietitian will be available to provide continuous support through a secure messaging app.

While in the dietary intervention phase of the study, participants will come to the UF Clinical and Translational Science Building once a week for 6 weeks. The study team will measure participant blood pressure and weight at each visit. At the first, middle, and final visits, the study team will collect a blood sample and urine sample from participants for lab testing, and participants will complete a short series of tests that measure physical performance.

Our ultimate research goal is to determine the effects of KD on body composition and clinically relevant measures of bone health and muscle function, as those data are needed to (1) inform the benefit-risk assessment for an older patient who is considering longer term adherence to KD therapy and (2) optimize the effectiveness of KD for age-related conditions.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* BMI 20 to <40 kg/m2
* Weight stable for last 12 months
* Male or female biological sex
* Willing to eat supplied food and adhere to dietary advice
* Willing to document food intake
* Willing to maintain weight
* Willing to attend study visits
* Smartphone ownership
* Community-dwelling with permanent living arrangement
* Resides within 30 miles of Gainesville, FL
* Willing to avoid alcohol intake
* Estimated energy requirement ≤ 2,700 kcal/day
* Have a refrigerator and means to reheat food within dwelling
* Bone mineral density tested within past 5 years or U.S. ethnicity-specific fracture risk assessment tool (FRAX) indicates ten year-probability of hip fracture <3% and ten year-probability of major osteoporotic fracture <20%

Exclusion Criteria:

* Pre- or peri-menopausal
* Fracture in past 6 months
* Circulating 25-hydroxyvitamin D < 20 ng/mL at screening
* History or prevalence of metabolic bone disease
* Chronic kidney disease diagnosis or eGFR <60 mL/min/1.73 m2 at screening
* Current or history of cancer excluding non-melanoma skin cancer
* Clinical cardiovascular disease, excluding current use of anti-hypertensive medication
* LDL cholesterol at screening that is elevated (≥ 160 mg/dL) or uncontrolled (≥ 100 mg/dL despise current statin treatment)
* History of recurrent kidney stones
* Current diabetes diagnosis
* Liver disease
* Pancreatic disease
* Heavy drinking per CDC definition
* Currently smoke tobacco
* Malabsorption disease including celiac and inflammatory bowel disease
* Inborn error of metabolism including disorders of fatty acid transport or oxidation, organic aciduria, porphyria, or familial hyperlipidemia
* Dementia diagnosis
* Dietary restrictions including food allergy, vegetarianism, veganism or gluten, dairy, or seafood avoidance
* Current or history of diagnosed eating disorder
* Thyroid disorder
* Male hypogonadism
* Menopause before age 40 years
* Gender-affirming hormone therapy
* Currently eat a ketogenic or Mediterranean diet based on ASA 24-hour dietary recall and Mediterranean diet screener
* Participation in concurrent research study
* Currently homeless
* Presence or possibility of co-morbid condition discovered during medical screening that would elicit safety concerns
* Living in skilled nursing facility
* Current gallbladder disease including gallstones
* History of 2 or more abdominal surgeries
* Current chronic constipation
* Current chronic diarrhea

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Rate of enrollment | Monthly. Up to 24 months.
  Number of participants enrolled in dietary intervention phase per month
Screen failure rate (percentage) | Monthly. Up to 24 months.
  Number of participants deemed ineligible / number of participants screened * 100
Treatment-specific retention rates | Either after the endline visit or when participant is withdrawn or withdraws from study
  Percentage of participants enrolled in dietary intervention phase who complete at least 6 intervention study visits including baseline, middle, and final visit.

SECONDARY OUTCOMES:
Treatment-specific adherence rates | Either after the endline visit or when participant is withdrawn or withdraws from study
  Treatment-specific adherence rates to protocol as evidenced by (1) dietary intake (2) blood ketone concentrations

OTHER OUTCOMES:
Bone turnover markers | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Serum CTX, urine NTX, serum TRACP-5b, serum P1NP, serum BSAP, serum osteocalcin
Body fat percentage | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Body Fat Percentage measured by dual-energy x-ray absorptiometry
Fat mass index | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Fat Mass Index measured by dual-energy x-ray absorptiometry
Visceral Adipose Tissue | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Visceral Adipose Tissue (VAT) measured by dual-energy x-ray absorptiometry
Fat Free Mass Index | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Fat Free Mass Index measured by dual-energy x-ray absorptiometry
Skeletal Muscle Mass | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Skeletal Muscle Mass measured by dual-energy x-ray absorptiometry
Appendicular Lean Mass to Height Ratio | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Appendicular Lean Mass to Height Ratio measured by dual-energy x-ray absorptiometry
Predicted resting metabolic rate | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Resting Metabolic Rate estimated from dual-energy x-ray absorptiometry data
24-hour urine analytes | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  A standardized report from 24-hour urine studies
Handgrip strength | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Handgrip strength measured by dynamometer
Total balance test score | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Results of balance tests performed as part of the short physical performance battery
Gait speed test score | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Results of gait speed tests performed as part of the short physical performance battery
Chair stand test score | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Results of chair stand tests performed as part of the short physical performance battery
Circadian clock gene expression | Pre-intervention; during the intervention (at 6 weeks into the intervention)
  Relative expression of circadian genes in whole blood collected in PAXgene blood RNA tubes
Vitamin D status | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Circulating concentrations of vitamin D metabolites
Circulating parathyroid hormone (PTH) concentration | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Circulating concentration of parathyroid hormone
Anion gap | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Anion gap from comprehensive metabolic panel
Insulin | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Circulating insulin concentration
Glucagon | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Circulating glucagon concentration
IGF-1 | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Circulating IGF-1 concentration
Beta-hydroxybutyrate | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Circulating beta-hydroxybutyrate concentration
Blood lipids | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Total Cholesterol, Triglycerides, HDL Cholesterol, LDL-Cholesterol, Non-HDL Cholesterol
Cystatin C | Pre-intervention; during the intervention (at 3 and 6 weeks into the intervention)
  Serum cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: Cora Best, PhD, RDN, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Available indefinitely after 3 years following study completion
Access Criteria: Reasonable request

DOCUMENTS (1):
  • Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT06203392/ICF_000.pdf